CLINICAL TRIAL: NCT03641144
Title: Navigation Laser Versus Traditional Laser Photocoagulation for Mild Diabetic Macular Edema：A Prospective, Randomized, Paralleled Clinical Trial
Brief Title: Navigation Laser Versus Traditional Laser Photocoagulation for Mild Diabetic Macular Edema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Chen-jin, Professor，Dr, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NLPD-ZOC
Record Dates: First submitted 2018-08-07; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; navigation laser; laser photocoagulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Navigation laser (Experimental): Navigation laser photocoagulation treatment to the macular area of retinal thickening with a focal pattern and/or grid pattern
  Interventions: Device: Navigation laser
- Traditional laser (Active Comparator): Traditional laser photocoagulation treatment to the macular area of retinal thickening with a focal pattern and/or grid pattern
  Interventions: Device: Traditional laser

INTERVENTIONS:
Device: Navigation laser — Navigation laser device is a scanning slit-based instrument.before treatment the surgeon plan laser spots on the screen based on image(infrared, colour, fluorescein angiography)and then apply automated patterns and single spots as appropriate.the device will automatically carry out the plan.
  Other Names: Navigation laser photocoagulation treatment
  Arms: Navigation laser
Device: Traditional laser — Traditional laser is a slitlamp based instrument.Surgeon operate traditional laer device while watching Participant's image(infrared, colour, fluorescein angiography) and then manually aim at and trigger laser.
  Other Names: Traditional laser photocoagulation treatment
  Arms: Traditional laser

SUMMARY:
The aim of this study is to evaluate treatment effect and safety of navigation laser photocoagulation for mild diabetic macular edema compared with traditional laser.

DETAILED DESCRIPTION:
navigation laser is a novel fundus imaging and laser treatment method that allows imaging (infrared, colour, fluorescein angiography) and integrated laser treatment of the retina. Besides documentation, precision,safety and patient comfort,the main theoretical advantages lie in retina navigation.This randomized, parallel controlled, clinical-trial aims to evaluate treatment effect and safety of navigation laser photocoagulation for mild diabetic macular edema compared with traditional laser. The primary outcome measures is the Best-corrected visual acuity (BCVA) of the participants at 1 year after treatment. Besides, the slit-lamp examination, tonometry, funduscopy, and OCT, FFA, ICGA examinations will also be compared between different groups to find the advantage of navigation laser .

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Diagnosed as diabetic retinopathy with Mild macular edema
* BCVA≥0.5
* No macular laser coagulation or surgery or medicine therapy of macular edema within the last 6 months

Exclusion Criteria:

* Blood glucose was not controlled steadily(HbA1cd≥10%)
* Accompanied with severe hypertension（BP≥180/110mmHg）
* Taking part in other clinical trial within 3 months
* Planning panretinal photocoagulation(PRP) within 3 months
* Performed cataract surgery in the last 3 months
* Accompanied with other retinal vascular disease that can lead to macular edema, for example branch retinal vein occlusion(BRVO),central retinal vein occlusion(CRVO)
* Accompanied with severe opacity of refractive media that maybe impact therapy and observation
* Accompanied with nystagmus
* Accompanied with some history that maybe interfere with result or increase the risk of patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity | 12 months
  Best Corrected Visual Acuity will be measured by standard Early Treatment Diabetic Retinopathy Study (ETDRS) protocol

SECONDARY OUTCOMES:
Central Retinal Thickness | 12 months
  Central Retinal Thickness will be performed by optical coherence tomography(OCT)
10°retinal sensitivity | 12 months
  Retinal sensitivity will be measured by microperimetry
treatment time | 1 hour
  treatment time is time from laser treatment beginning to end
Participants pain intensity | 1 hour
  Participants pain intensity will be immediately measured by Visual Analogue Scale/Score （VAS）after treatment.The VAS is a straight horizontal line of fixed length（100 mm）. The ends are defined as the extreme limits of the parameter to be measured (pain) orientated from the left (0) to the right (100).The patient marks on the line the point that participants feel represents their perception of their current pain intensity.the VAS score is determined by measuring the distance (mm) on the 100mm line between the "0" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm) .
Number of laser spots within macular fovea | 1 month
  Number of laser spots within macular fovea will measured by foundus photograph

CONTACTS AND LOCATIONS:
Overall Officials: Chenjin Jin, Ph.D, Study Chair — State Key Laboratory of Ophthalmology, Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided